CLINICAL TRIAL: NCT02783391
Title: Pre and Per-operative Electrophysiological Cartography of Speech Area With Cortical Electrode Matrices
Acronym: BRAINSPEAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRAINSPEAK
Record Dates: First submitted 2016-05-12; First posted 2016-05-26 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Tumoral or Epileptical Cortectomy
MeSH Terms: interventions — Electrocorticography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BRAINSPEAK (Experimental): Electrocorticographical (ECoG) and intracortical electrodes
  Interventions: Device: ECoG and intracortical electrodes

INTERVENTIONS:
Device: ECoG and intracortical electrodes

SUMMARY:
New method for speech area cartography in patient individual cortical anatomy in view of improving functional area limit preservation during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing cortectomy
* Male or female aged over 18 years
* Registered in the French social security scheme
* Signed informed consent

Exclusion Criteria:

•All categories of protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
electrophysiological recording | 2 hours
  Electrophysiological recording of brain Speech Area, using Cortical Electrode Matrices, in order to improve functional area limit preservation during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No